CLINICAL TRIAL: NCT07364123
Title: Education and Telephone Counseling to Improve Adherence to Immunosuppressive Medication in Kidney Transplant Recipients: A Randomized Controlled Trial
Brief Title: Kidney Transplant Immunosuppressive Therapy Adherence Trial (KITE)
Acronym: KITE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Tuğba Albayram, Research Assistant Dr, University of Gaziantep
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022/441
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Kidney Transplantation; Medication Non-Adherence; Immunosuppressive Therapy; Renal Transplant Recipients
Keywords: Kidney Transplant; Immunosuppressive Medication; Medication Adherence; Telephone Counseling; Patient Education; Tacrolimus Levels
MeSH Terms: conditions — Medication Adherence | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either an education plus telephone counseling group or a standard care control group, and both groups will be followed over 8 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education and Telephone Counseling Program (Experimental): A nurse-led structured education session covering immunosuppressive medication use, side effects, timing, and self-management strategies. Participants receive an educational booklet and are provided with scheduled telephone counseling sessions designed to reinforce adherence, address patient questions, and support problem-solving. All calls and follow-up interactions are documented. Pre-test, post-test, and follow-up adherence assessments are administered.
  Interventions: Behavioral: Education and Telephone Counseling Program
- Standart Care (No Intervention): Participants receive standard post-transplant clinical follow-up provided by the hospital, without additional structured education or telephone counseling. Routine care includes medical assessments and medication management per standard transplant center procedures.

INTERVENTIONS:
Behavioral: Education and Telephone Counseling Program — A nurse-led structured behavioral intervention designed to improve adherence to immunosuppressive medication. The intervention includes an individualized education session at discharge, provision of an educational booklet, and scheduled telephone counseling at 7-15 days, 4 weeks, and 8 weeks. Participants also receive access to a dedicated phone line for additional support. Counseling focuses on medication routines, problem-solving strategies, reinforcing adherence behaviors, and addressing patient concerns. Pre-test and post-test assessments are used to evaluate changes in knowledge and adherence.
  Other Names: Immunosuppressive Adherence Education; Nurse-Led Tele-Counseling
  Arms: Education and Telephone Counseling Program

SUMMARY:
This randomized controlled interventional study aims to evaluate the effect of structured education and telephone counseling on immunosuppressive medication adherence among kidney transplant recipients. Poor adherence to immunosuppressive therapy after kidney transplantation is a major risk factor for acute rejection, graft loss, and increased morbidity. Education and behavioral support interventions delivered by nurses may improve medication understanding, adherence behaviors, and self-management skills.

In this trial, 60 participants will be randomly assigned to either an intervention group receiving individualized education, an immunosuppressive medication adherence booklet, and scheduled telephone counseling sessions, or a control group receiving routine clinical care. Adherence will be assessed using the Immunosuppressive Medication Adherence Scale and biological monitoring through tacrolimus level variability over 8 weeks. Additional outcomes include changes in medication knowledge scores based on pre-test and post-test assessments.

The study will contribute evidence regarding whether nurse-led telephone counseling and structured education can enhance adherence, improve clinical follow-up, and support long-term graft success in kidney transplant patients.

DETAILED DESCRIPTION:
Kidney transplant recipients are required to follow lifelong immunosuppressive therapy to prevent rejection and preserve graft function. However, studies consistently demonstrate substantial rates of non-adherence, which is associated with increased acute rejection, graft dysfunction, hospitalization, and higher long-term mortality. Behavioral, educational, and psychosocial factors play critical roles in medication adherence, particularly during the early post-transplant period when patients must adapt to complex medication regimens and lifestyle changes.

This randomized controlled trial was designed to evaluate whether a structured nurse-led education program combined with scheduled telephone counseling can improve adherence to immunosuppressive medication among kidney transplant recipients. The intervention includes individualized education, distribution of an adherence-focused patient booklet, reinforcement of medication-taking routines, problem-solving support, and ongoing telephone follow-up to address questions and encourage self-management behaviors.

Participants are randomly assigned to an intervention group or a usual-care control group. Adherence is assessed using a validated self-report scale and by monitoring variability in tacrolimus levels, which is commonly used as an objective indicator of medication-taking consistency. The assessment schedule includes baseline and follow-up evaluations over 8 weeks. The study also incorporates pre-test and post-test evaluations to measure changes in participants' medication knowledge following the educational intervention.

The results of this study are expected to provide evidence on whether integrating telehealth-based nursing support into routine post-transplant care improves medication adherence and supports better clinical outcomes. The intervention model developed here may offer a practical, patient-centered strategy that can be adopted in transplant centers with limited resources.

ELIGIBILITY:
Inclusion Criteria:

* Adult kidney transplant recipients aged 18 years or older
* At least 1 month post-kidney transplantation
* Able to provide informed consent
* Cognitively intact and oriented to person, place, and time
* Able to communicate via telephone
* Voluntarily willing to participate in the study

Exclusion Criteria:

* Under 18 years of age
* Severe cognitive impairment preventing participation
* Inability to communicate effectively (hearing or speech limitations without support)
* Patients who do not meet the post-transplant time threshold (less than 1 month)
* Patients unwilling or unable to participate in follow-up sessions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Adherence Score to Immunosuppressive Medication | Baseline and Week 8
  Medication adherence will be assessed using the Immunosuppressive Medication Adherence Scale (11 items). Total scores range from 11 to 55, with higher scores indicating better medication adherence. Participants will complete the scale at baseline and at Week 8. An increase in score reflects improved adherence following the education and telephone counseling intervention.

SECONDARY OUTCOMES:
Variability in Tacrolimus Trough Levels | Baseline and Week 8
  Tacrolimus trough concentrations will be monitored during routine clinical visits. Variability will be calculated using the standard deviation (SD) of trough levels between baseline and Week 8. An SD greater than 2.48 is considered indicative of medication non-adherence according to predefined clinical criteria. Lower variability reflects better biological consistency of medication adherence.
Medication Knowledge Score | Medication knowledge will be assessed using a 22-item questionnaire on dosage, timing, side effects, interactions, and rejection signs. Scores range 0-22; higher scores indicate better knowledge. Assessed at baseline, Week 4, and Week 8.
  4 weeks and 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziantep University Sahinbey Research and Application Hospital, Gaziantep, Şehitkamil, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual patient data (IPD) will not be shared because the dataset contains sensitive clinical information, including laboratory values and medication adherence details from kidney transplant recipients. Due to privacy concerns, ethical considerations, and institutional regulations regarding the protection of personal health data, de-identified datasets will not be made publicly available. Aggregated results will be reported in publications without revealing individual-level data.

REFERENCES:
- [Background] 1. De Bleser, L., Dobbels, F., Berben, L., Vanhaecke, J., Verleden, G. ve diğerleri. (2011). The Spectrum of Nonadherence with Medication in Heart, Liver, and Lung Transplant Patients Assessed in Various Ways. Transplant International, 24, 882-891. 2. Denhaerynck, K., Dobbels, F., Cleemput, I., Desmyttere, A., Keller, PS. ve diğerleri. (2005). Prevalence, Consequences and Determinants of Nonadherence in Adult Renal Transplant Patients: a literatüre review. Transplant International, 18, 1121-1133. 3. Dew, MA., Di Martini, AF., De Vito Dabbs, A., Myaskovsky, L. ve diğerleri. (2007). Rates and Risk Factors for Nonadherence to the Medical Regimen After Adult Solid Organ Transplantation. Transplantation, 83, 858-873. 4. Hansen, R., Seifeldin, R. ve Noe, L. (2007). Medication Adherence in Chronic Disease: Issues in Posttransplant Immunosuppression. Transplantation Proceedings, 39, 1287-1300. 5. Vlaminck, H., Maes, B., Evers, G., Verbeke, G. ve Lerut, E. (2004). Prospectives Study on Late Consequences of Subclinical Non-Compliance with Immunosuppressive Therapy in Renal Transplant Patients. American Journal of Transplantation, 4, 1509-1513. 6. Butler, J.A., Roderick, P., Mullee, M., Mason J.C. ve Peveler R.C. (2004). Frequency and Impact of Nonadherence to Immunosuppressants After Renal Transplantation: A Systematic Review. Transplantation, 77(5), 769-776. 7. Dobbels, F., De Geest, S. ve Van Cleemput, J. (2004). Effect of Late Medication Non-Compliance on Outcome After Heart Transplantation: a 5 Year Follow-Up. Journal of Heart and Lung Transplantation, 23, 1245. 8. Morrissey, P.E., Reinert, S., Yango, A., Gautam, A., Monaco A. ve Gohh R. (2005). Factors contributing to acute rejection in renal transplantation: the role of noncompliance. Transplant Proceedings, 37(5), 2044-2047. 9. Michelon, T.F., Piovesan, F., Pozza, R., Castilho, C., Bittar, A.E., Keitel, E. ve diğerleri. (2002). Noncompliance as a Cause of Renal Greft Loss. Transplantation Proceeding, 34(7), 2768-2770.